CLINICAL TRIAL: NCT02694926
Title: National (German-wide) Education Programme for Patients With Chronic Adrenal Insufficiency
Brief Title: National Education Programme for Patients With Chronic Adrenal Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Dr. Michael Droste, Elisenstraße 12, 26122 Oldenburg (Unknown); Prof. Dr. Marcus Quinkler, Praxis für Endokrinologie,10627 Berlin (Unknown); Dr. Gesine Meyer, Universitätsklinikum Frankfurt, 60590 Frankfurt am Main (Unknown); PD Dr. Nicole Reisch, LMU München, D-80336 München (Unknown); Prof. Dr. Holger Willenberg, Zentrum für Innere Medizin, D-18057 Rostock (Unknown); Prof. Johannes Klein, Zentrum Endokrine Medizin, 23564 Lübeck (Unknown); Charite University, Berlin, Germany (Other); MVZ Endokrinologikum Saarbrücken, Europaallee 15, 66113 Saarbrücken (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Nationales Schulungsprogramm
Record Dates: First submitted 2016-02-08; First posted 2016-03-01 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Adrenal Insufficiency
Keywords: adrenal crisis; education programme
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adrenal insufficiency (Other)
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — During a session of 90 minutes duration, patients are educated in basic knowledge on adrenal insufficiency including the correct behaviour in emergency settings.

SUMMARY:
Even under established replacement therapy, patients with adrenal insufficiency still suffer from impaired quality of life and experience adrenal crises. Patient education is regarded as important preventive measure. In this study a german-wide standardized education Programme will be evaluated.

DETAILED DESCRIPTION:
Design aspects:

In a prospective trial the efficiency of a german-wide education programme in patients with chronic adrenal insufficiency will be evaluated by using a questionnaire before and after training.

Patients:

Patients will be recruited out of the patient population of the participating nine medical centers. To achieve a anticipated number of 450 patients, each center will include al least 50 patients with chronic adrenal insufficiency under established replacement therapy .

Trial flow:

During sessions of 90 minutes duration, patients and relatives are educated in basic knowledge on adrenal insufficiency including the correct behaviour in emergency settings. Participants are provided with emergency cards and sets and are trained in self-injection of glucocorticoids. To evaluate the standardized education programme, patients complete three questionnaires (before, shortly after and 6-9 months after the training) at nine endocrine centres. All centres had been certified by the German Endocrine Society for the education programme. Questionnaires assess general knowledge on adrenal insufficiency and document the influence on patients' feeling of security.

Statistical Analysis:

Documentation and analysis will be performed at the Department of Medicine I, Endocrine and Diabetes Unit, University of Würzburg, Germany. Data will be documented after pseudonymisation in a data base. Data analysis is mainly descriptive.

Stopping rules:

Participation of patients is fully voluntarily. Patients are able to stop participation in the study at any point in time. In addition, patients might claim the elimination of all data material at any point in time.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* patient's written informed consent
* Ability to comply with the protocol procedures
* patients with primary or secondary adrenal insufficiency under established stable replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2014-12; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Efficiency of education evaluated by questionnaire. | 12-24 months
  To evaluate the efficiency of the education programme patients complete three questionnaires. Questionnaires asses the general knowledge on adrenal insufficiency and the correct behavior in emergency settings via multiple choice questions. Overall scores before and after training will be compared

SECONDARY OUTCOMES:
Patient satisfaction /safety evaluated by questionnaire. | 12-24 months
  Evaluation via questionnaire including subjective multiple choice questions e.g. on the feeling of safety.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Hahner, MD, Prof., Principal Investigator — University Hospital Wuerzburg
Locations (1):
- University Hospital Wuerzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
publication of collected data in medical journals and specialist congresses

REFERENCES:
- [Background] Hahner S, Spinnler C, Fassnacht M, Burger-Stritt S, Lang K, Milovanovic D, Beuschlein F, Willenberg HS, Quinkler M, Allolio B. High incidence of adrenal crisis in educated patients with chronic adrenal insufficiency: a prospective study. J Clin Endocrinol Metab. 2015 Feb;100(2):407-16. doi: 10.1210/jc.2014-3191. Epub 2014 Nov 24. PMID 25419882
- [Background] Hahner S, Hemmelmann N, Quinkler M, Beuschlein F, Spinnler C, Allolio B. Timelines in the management of adrenal crisis - targets, limits and reality. Clin Endocrinol (Oxf). 2015 Apr;82(4):497-502. doi: 10.1111/cen.12609. Epub 2014 Nov 6. PMID 25200922
- [Background] Hahner S, Loeffler M, Bleicken B, Drechsler C, Milovanovic D, Fassnacht M, Ventz M, Quinkler M, Allolio B. Epidemiology of adrenal crisis in chronic adrenal insufficiency: the need for new prevention strategies. Eur J Endocrinol. 2010 Mar;162(3):597-602. doi: 10.1530/EJE-09-0884. Epub 2009 Dec 2. PMID 19955259
- [Background] Allolio B. Extensive expertise in endocrinology. Adrenal crisis. Eur J Endocrinol. 2015 Mar;172(3):R115-24. doi: 10.1530/EJE-14-0824. Epub 2014 Oct 6. PMID 25288693
- [Background] Smans LC, Van der Valk ES, Hermus AR, Zelissen PM. Incidence of adrenal crisis in patients with adrenal insufficiency. Clin Endocrinol (Oxf). 2016 Jan;84(1):17-22. doi: 10.1111/cen.12865. Epub 2015 Aug 27. PMID 26208266
- [Background] Reisch N, Willige M, Kohn D, Schwarz HP, Allolio B, Reincke M, Quinkler M, Hahner S, Beuschlein F. Frequency and causes of adrenal crises over lifetime in patients with 21-hydroxylase deficiency. Eur J Endocrinol. 2012 Jul;167(1):35-42. doi: 10.1530/EJE-12-0161. Epub 2012 Apr 18. PMID 22513882
- [Background] Repping-Wuts HJ, Stikkelbroeck NM, Noordzij A, Kerstens M, Hermus AR. A glucocorticoid education group meeting: an effective strategy for improving self-management to prevent adrenal crisis. Eur J Endocrinol. 2013 May 17;169(1):17-22. doi: 10.1530/EJE-12-1094. Print 2013 Jul. PMID 23636446
- See also: German society of endocrinology — http://www.endokrinologie.net/